CLINICAL TRIAL: NCT01209897
Title: Testing Alternative Stage Models of Smoking Cessation: An Intervention Study
Brief Title: Testing Different Theories of Smoking Cessation: An Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Thaddeus Herzog, Principal Investigator, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA120799-02 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-09-27 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation
Keywords: Smoking
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stage of Change (Active Comparator): Participant received booklet based on stage of change.
  Interventions: Behavioral: Smoking cessation booklet
- Common Sense Model (Experimental): Participant received booklet based on common sense model.
  Interventions: Behavioral: Smoking cessation booklet
- Action Model (Active Comparator): Participant received booklet based on the action stage of change.
  Interventions: Behavioral: Smoking cessation booklet

INTERVENTIONS:
Behavioral: Smoking cessation booklet

SUMMARY:
The topic of this research is cigarette smoking cessation. We designed four smoking cessation booklets. These booklets are designed for smokers who differ in their motivation to quit smoking. We will compare different ways of matching booklets to smokers who vary in their motivation to quit smoking.

DETAILED DESCRIPTION:
The topic of the proposed research is adult cigarette smoking cessation. The PI has designed a set of four smoking cessation booklets. These booklets cover different aspects of the smoking cessation process, and are designed to help smokers who differ in their levels of motivation to quit smoking. The purpose of the study is to compare different ways of matching booklets to smokers who vary in their motivation to quit smoking. Adult smokers (N=1,826) will be recruited via newspaper ads, fliers, and possibly other methods, depending on response rates. Participants will enroll in the study by telephoning the research staff in response to the advertisements. The smoking cessation booklets and surveys will be sent via US Mail. Smokers will be assigned randomly to one of three intervention conditions. Participants at baseline will answer a series of survey items regarding their motivation and plans (or lack thereof) for quitting smoking. The three intervention conditions differ in that each employs a different method of matching smokers to one of the four booklets. Essentially, we are comparing different strategies for allocating booklets to smokers. Participants will be surveyed two weeks and two months after receiving their smoking cessation booklet.

ELIGIBILITY:
Inclusion Criteria:

* must be a current smoker who smokes at least three cigarettes per day
* must have smoked at least 100 cigarettes in their lifetime.
* must be able to read English so that they can read the intervention booklets and complete questionnaires in English.
* must have a mailing address so that they can receive booklets and questionnaires in the mail.
* must be age 18 or older.
* must live in Hawaii

Exclusion Criteria:

* not a current smoker
* smokes fewer than three cigarettes per day
* has not smoked at least 100 cigarettes in their lifetime
* cannot read English
* has no mailing address
* is under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1826 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Smoking Status | two months
  Participants will be asked if they are still smoking cigarettes, or if they have ceased to smoke cigarettes.

SECONDARY OUTCOMES:
Motivation to quit smoking | two months
  Participants will be asked about the extent to which they are motivated to quit smoking (for example, if they intend to quit smoking or do not intend to quit smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus A Herzog, Ph. D., Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States